CLINICAL TRIAL: NCT00668252
Title: Impact of Endogenous Sexual Hormones (Oestrogens and Testosterone) on the Endothelium Circulatory on Rolling at the Young and Old Healthy Volunteer.
Brief Title: Circulating Endothelium Progenitor Cells and Endogenous Oestrogen in Healthy Subjects
Acronym: Oestropec
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Yannick Vacher, Department Clinical Research of Developpement
Other Study IDs: P050904
Record Dates: First submitted 2008-04-09; First posted 2008-04-29 (Estimated); Last update posted 2008-04-29 (Estimated); Status verified 2006-03

CONDITIONS: Healthy
Keywords: endothelial progenitor cells; estrogen; menopause; cardiovascular risk

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — whole peripheral blood (150 ml)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Non menopausal women
- 2: age matched men
- 3: Menopausal women
- 4: age matched men

SUMMARY:
The purpose of this study is to determine whether the number of circulating EPC is different between healthy women and men.

DETAILED DESCRIPTION:
Study design: Open pilot study in health volunteers in the Hospital Saint-ANTOINE's Clinical Investigation Centre (CIC).

Recruitment and course of the study: The subjects will be recruited among the CIC's pool of healthy volunteers. Volunteer people will then have biological and clinical baseline examinations. If they match the inclusion criteria, an appointment will be taken for the blood sample intend for the characterization of the EPC and hormonal plasma levels evaluation. The participation will not exceed 2 months. Young women will have to come between the 9th and the 11th day after the beginning of menses). A total of 150 ml of peripheral blood will be collected. The study will last 18 months.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 19 and 25 kg/m²
* non menopausal women :
* age 18 to 40 years,
* regular menstrual cycles
* no hormone therapy as contraceptives
* postmenopausal women :
* age above 55 years old
* amenorrhoea since 5 years at least
* no hormone therapy since at least 3 month

Exclusion Criteria:

* no medical insurance
* inclusion in another study
* smoking, Statins treatment, uncontrolled diabetes or hypertension and personal history of cardiovascular disease.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2006-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Number of endothelial progenitor cells by cytometry | Baseline

SECONDARY OUTCOMES:
To compare the number of EPC in young women to older men and menopausal women. To evaluate the correlation between the number of EPC and 17 b-estradiol plasma level. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Tabassome Simon, MD - PhD, Principal Investigator — Assistance Publique Hopitaux de Paris - Université Pierre et Marie Curie Paris 6
Locations (1):
- Assistance Publique Hopitaux de Paris - Hopital Saint Antoine, Paris, France